CLINICAL TRIAL: NCT03954925
Title: Anatomic Anterior Cruciate Ligament With Short Hamstring Graft Compare With a Standard Hamstring Graft Technique: Prospective Cohort Study
Brief Title: Anatomic Anterior Cruciate Ligament With Short Hamstring Graft Compare With a Standard Hamstring Graft Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Collaborators: Thammasat University (Other)
Responsible Party: Principal Investigator, Jatupon Kongtharvonskul, principle investigator, Ramathibodi Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTU-EC-OT-0-255-61
Record Dates: First submitted 2019-05-13; First posted 2019-05-17 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: ACL; short hamstring graft; standard hamstring graft
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anatomic anterior cruciate ligament with short hamstring (Active Comparator): Anatomic anterior cruciate ligament with short hamstring graft
  Interventions: Procedure: Anatomic anterior cruciate ligament with short hamstring graft technique
- Anatomic anterior cruciate ligament with standard hamstring (Active Comparator): Anatomic anterior cruciate ligament with standard hamstring graft
  Interventions: Procedure: Anatomic anterior cruciate ligament with a standard hamstring graft technique

INTERVENTIONS:
Procedure: Anatomic anterior cruciate ligament with short hamstring graft technique — ACL and short hamstring graft
  Arms: Anatomic anterior cruciate ligament with short hamstring
Procedure: Anatomic anterior cruciate ligament with a standard hamstring graft technique — ACL with standard hamstring graft
  Arms: Anatomic anterior cruciate ligament with standard hamstring

SUMMARY:
this study was to evaluate the functional outcome of quadruple hamstring graft in femoral tunnel less than 15 mm and morethan or equal 15 mm of ACL reconstruction. The hypothesize that no difference intermediate follow up ( 6 month - 24 month) of functional outcome and clinical evaluation between short and normal femoral tunnel graft length of hamstring tendon ACL reconstruction.

DETAILED DESCRIPTION:
The patient recruitment (N=29) and baseline data collection were done at our institute between March2014-September 2015. The inclusion criteria were patients with anterior cruciate ligamentous injury who needed ligamentous reconstruction, closed growth plates and younger than 60 years old, absence of ligament injury to the opposite knee. The exclusion criteria are patients who did not want to participate in this study or patient with failed anterior cruciate ligamentous reconstruction.

All the procedure of anterior cruciate ligament reconstructions were performed by the senior authors (B.C). Semitendinosus and gracilis tendons were harvested through an oblique approach medial to the tibial tubercle in all patients. Complete anterior cruciate ligament was confirmed at arthroscopy. Associated intra-articular injuries such as meniscus tear and cartilage lesions were fixed at of the index operation .The femoral tunnel were drilled though the AM portal.

ELIGIBILITY:
Inclusion Criteria:

* Patients with anterior cruciate ligamentous injury with the diagnosis of injured ligaments was made based on a detailed history of the knee injury, physical examination on pathologic status and abnormal laxity, routinely performed plain radiographs and MRI scans, and the findings at surgery.
* Patients who have closed growth plates.
* Patients who younger than 60 years old.
* Patients who absence of ligament injury to the opposite knee.

Exclusion Criteria:

* Patients with a combined ligament injury as folling:

  1. Posterior cruciate ligament
  2. The lateral collateral ligament
  3. The posterolateral corner structures of the knee
  4. Medial collateral ligament.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Visual analog score | 18 months
  visual analog score rang from 0-10 (minimum=0, maximun=10) and the higher values represent a worse outcome?)

SECONDARY OUTCOMES:
range of motion | 18 months
  range of motion range from 0-160 degree and the higher values represent a better outcome
complication | 18 months
  number of participant who have infection, stiffness and re-operation

IPD SHARING:
Plan to Share IPD: No